CLINICAL TRIAL: NCT06301568
Title: Retrospective Analysis of Long-term Speech Performance in Cochlear Implant Recipients Using Electro-acoustic Stimulation
Status: Recruiting | Type: Observational
Sponsor: Advanced Bionics AG (Industry)
Responsible Party: Sponsor
Other Study IDs: ABIntl-23-12
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Cochlear Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective study designed to collect long-term speech perception results for cochlear implants recipients using electro-acoustic-stimulation as measured in the clinical routine and to confirm the performance of sound processors associated with acoustic earhooks.

ELIGIBILITY:
Inclusion Criteria:

* Being implanted with HiRes Ultra or HiRes Ultra 3D SlimJ
* Being a user of the "acoustic earhook" system
* Having provided informed consent regarding use of his/her data for research.

Exclusion Criteria:

* no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The studied population consists of all CI users implanted with a HiRes Ultra or HiRes Ultra 3D SlimJ between January 2017 and August 2022 and using an acoustic earhook at the Medical University of Hannover in Germany (MHH)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Freiburger monosyllabic word recognition score in quiet | 12 months after device activation
  Percent correct in the Freiburger Monosyllabic Word test

SECONDARY OUTCOMES:
HSM sentence score or OlSa recognition score in quiet | 12 months after device activation
  percent correct in either the HSM sentence test or the Oldenburger sentence test

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Büchner, Principal Investigator — Hannover Medical School
Locations (1):
- Medizinische Hochschule Hannover, Hanover, Germany